CLINICAL TRIAL: NCT02533024
Title: Preoperative Prevalence of Ulnar Neuropathy and Changes in Ulnar Nerve Latency During Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ulnar-Neuropathy-ULE
Record Dates: First submitted 2015-08-20; First posted 2015-08-26 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2016-09

CONDITIONS: Ulnar Neuropathy
MeSH Terms: conditions — Ulnar Neuropathies | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group Cohort (Experimental): All subjects will have nerve conduction studies (Electromyography/EMG) pre-operatively, monitored intra-operatively and immediately post-operative.
  Interventions: Other: Electromyography

INTERVENTIONS:
Other: Electromyography — All subjects will have an EMG before, during and immediately after surgery.
  Other Names: EMG

SUMMARY:
This study is to investigate the incidence of undiagnosed ulnar neuropathy in patients undergoing surgery. The investigators hope to determine if patients with ulnar neuropathy have changes in nerve conduction latency during surgery.

DETAILED DESCRIPTION:
After obtaining an informed consent, the participating subjects will be asked a few questions relating to ulnar nerve dysfunction. Following this the investigators will do a focused physical exam looking for decrement of sensation in the distribution of the ulnar nerve and muscle strength of the hand muscles supplied by the ulnar nerve. After this the subjects will undergo an EMG exam to measure the conduction velocity of the ulnar nerve. Basically the nerve will be stimulated with a small current and the resultant muscle activity of the hand muscle will be picked up using an EKG like patch applied to the skin over the hand. If a subject is diagnosed to have ulnar neuropathy preoperatively the investigators would study the EMG based nerve conduction during surgery at 30-60 minute intervals for the duration of surgery. For purposes of comparison the investigators would measure the ulnar nerve conduction during surgery in age and sex matched controls.

ELIGIBILITY:
Inclusion Criteria:

* 50 yrs of age or older
* Scheduled to undergo a surgical procedure at UTMC with an anticipated length of 2hours or greater

Exclusion Criteria:

* Less than 50yrs
* Not scheduled for a surgical procedure at UTMC or scheduled for a surgical procedure with an anticipated length of less than 2hours

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-08; Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of ulnar neuropathy in patients scheduled to undergo anesthesia and surgery as measured by electromyography | Day 1
  Prevalence of undiagnosed or subclinical ulnar neuropathy as determined by electromyography

SECONDARY OUTCOMES:
Amplitude (mV) | Day 1
  Compare preoperative, perioperative and postoperative amplitude changes from EMG
Latency (ms) | Day 1
  Compare preoperative, perioperative and postoperative latency changes from EMG
Velocity (m/s) | Day 1
  Compare preoperative, perioperative and postoperative velocity changes from EMG

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B Casabianca, MD, Principal Investigator — University of Toledo
Locations (1):
- University of Toledo, Toledo, Ohio, United States